CLINICAL TRIAL: NCT02774434
Title: Efficacy Study of the Draeger Jaundice Meter (JM-105) in Providing TcB Measurements to Estimate TSB in Neonates of ≥ 24 Weeks of Gestational Age Who Have and Have Not Undergone Phototherapy
Brief Title: Efficacy Study of the Draeger Jaundice Meter (JM-105) in Neonates of ≥ 24 Weeks of Gestational Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Draeger Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: JM-105 Study
Record Dates: First submitted 2016-05-06; First posted 2016-05-17 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Hyperbilirubinemia; Neonatal Jaundice
MeSH Terms: conditions — Hyperbilirubinemia; Jaundice, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- JM-105 (Experimental): Within 15 minutes of each ordered blood sample 2 TcB measurements will be performed using the JM-105 on the sternum and forehead. Subject's participation will end after a 10 day period.
  Interventions: Device: JM-105

INTERVENTIONS:
Device: JM-105 — Measurement of TcB via the JM-105 device

SUMMARY:
The Canadian Pediatric Society recently published guidelines to monitor bilirubin levels and as part of standard of care all hospitalized newborns are routinely monitored for the development of high bilirubin or jaundice every 8-12 hours. One device approved and used in both Canada and the United States is the Draeger Jaundice Meter JM-103, a non-invasive medical device. It has been proven to be effective in patients >35 weeks gestational age. Recently the JM-103 has been upgraded to include a bigger touch screen, greater storage and functionality. The rest of the features of the JM-103 and JM-105 are identical. In order to test the accuracy of the JM-105 neonates from ≥ 24 weeks gestational age who have or have not undergone phototherapy will be prospectively monitored for transcutaneous bilirubin (TcB) using the JM-105. The measurements will be compared to a physician-ordered total serum bilirubin (TSB).

DETAILED DESCRIPTION:
Hyperbilirubinemia is a condition that occurs in newborns when there is too much bilirubin in the blood. It is the most common cause of newborns being readmitted to the hospital. It may be harmless or harmful depending on what the cause is and how bad it is. The serum level of bilirubin required for jaundice varies with infants skin tones and body region, however jaundice usually becomes visible in the white part of the eye at smaller levels. Although jaundice in newborn is generally not harmful, it is important to monitor newborns to identify those that are at risk of developing a neurological dysfunction from high bilirubin levels. As part of standard of care all hospitalized newborns are routinely monitored for the development of jaundice by nursing staff and physicians every 8-12 hours. Although jaundice in newborns can usually be detected by lightening/whitening in the skin with digital pressure, this method of visual estimation is very inaccurate and unreliable. Transcutaneous bilirubin measurements are non-invasive and has proven to be equivalent to total serum bilirubin measurements. The JM-103 has been proven to be an effective TcB measure in ethnically diverse populations for patients >35 weeks gestational age. The JM-105 has been upgraded from the JM-103 with greater efficiency and accuracy. The basic function is the same but has been improved with a larger touch screen, data storage and transmission functionality.

This prospective multi-centre study will be conducted to determine the diagnostic accuracy and performance of the use of the JM-105 in providing transcutaneous bilirubin measurements to estimate serum total bilirubin in neonates ≥ 24 weeks of gestational age who have or have not undergone phototherapy. The study will compare each of the measurements of transcutaneous bilirubin (TcB) obtained for 10 days via the JM-105 device with a neonatology team-ordered series of serum total bilirubin (TSB) measured by high-performance liquid chromatography.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a neonate ≥24 weeks of gestational age for whom a course of phototherapy has not started, is in progress or has been completed
* The subject's routine management includes TSB evaluations
* The subject's family are willing and able to participate in baseline and TSB measurements over 10 days
* Written informed consent to participate in the study has been provided by the subject or legal representative (parent or legal guardian in a clinical study involving children)

Exclusion Criteria:

* The subject has Hydrops fetalis
* The subject has major congenital malformations, diseases or skin conditions or thickness that, in the opinion of the investigator would preclude or interfere with the use of the JM-105

Ages: 24 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 464 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Accuracy of TcB measured with the JM-105 device in predicting the Serum Bilirubin measurements performed on blood samples | Within 15 minutes of blood sample taking
  Primary objective is to determine the accuracy of TcB measured with the JM-105 device in predicting the Serum Bilirubin measurements performed on blood samples from heel sticks or from peripheral line in neonates ≥ 24 weeks of gestational Age who are currently undergoing or have undergone phototherapy as a Screening and Monitoring device for hyperbilirubinemia

SECONDARY OUTCOMES:
Normalized curve of TSB measurements using the JM-105 | Within 15 minutes of blood sample taking
  The secondary objective is to determine a normalized curve of TSB measurements using the JM-105.
Influence of phototherapy on TSB measurements | Within 15 minutes of blood sample taking
  The Impact of phototherapy on TSB measurements will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sgro, MD, Principal Investigator — Unity Health Toronto
Locations (3):
- Canada (3):
  - Saint Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Hamilton Health Science Centre, Toronto, Ontario

REFERENCES:
- [Derived] Jegathesan T, Campbell DM, Ray JG, Shah V, Berger H, Hayeems RZ, Sgro M; NeoHBC. Transcutaneous versus Total Serum Bilirubin Measurements in Preterm Infants. Neonatology. 2021;118(4):443-453. doi: 10.1159/000516648. Epub 2021 Jun 17. PMID 34139689